CLINICAL TRIAL: NCT00413842
Title: Effects of tDCS Over the Cerebellum on Motor Function
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070049; 07-N-0049
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-20

CONDITIONS: Healthy
Keywords: Transcranial Direct Current Stimulation (tDCS); Plasticity; Primary Motor Cortex; Cerebellum; Transcranial Magnetic Stimulation (TMS); Healthy Volunteer; HV

SUMMARY:
This study will evaluate whether applying electrical stimulation on the cerebellum (posterior and lower part of the brain) can influence brain excitability and hand movement performance.

A new technique became available to stimulate the brain: transcranial direct current stimulation (tDCS), which could improve the ability to learn. Researchers do not know whether applying tDCS over the cerebellum could also influence motor function, and they want to examine changes in brain excitability, by using transcranial magnetic stimulation (TMS).

Patients ages 18 to 40 who are not pregnant may be eligible for this study. They will come to NIH for a medical history and completing a questionnaire about memory and attention. There will be five experiments, each up to 5 hours, for about 1 to 5 weeks, in which patients perform tasks like pinching a special device between the thumb and index fingers, or reaching for target objects on the computer screen. Patients will receive mild electrical stimulation over a different part of the head each day. Some experiments are done without the electrical current, but patients will not know which ones are with or without stimulation. There are also short questionnaires about attention, fatigue, and mood, to be completed before, during, and after each experiment.

Patients will be connected to an electromyography (EMG) machine, to measure electrical activity of muscles. Electrodes are taped to the skin over one small hand muscle. TMS allows electrical pulses to pass through the brain to stimulate it. TMS is used at the beginning of each experiment to determine the precise location on the scalp of two target areas: cerebellum and motor cortex. TMS is a safe procedure. Discomfort, headache, or nausea can occur, but all symptoms usually go away promptly. During motor learning under tDCS, also a safe procedure, patients sit in a comfortable chair, and the arm and wrist and arm are kept still. Sponge electrodes are applied on the chin, back of the head, neck, collarbone, lateral part of the head, or above the eyebrow. A small electrical current is passed between electrodes. Patients may feel an itching or tingling sensation under the electrodes or see slight light flashes. tDCS is applied for 20 to 30 minutes. A magnetic resonance imaging (MRI) scan, which may also be involved, uses a strong magnetic field and radio waves to obtain images of body organs and tissues. Patients lie on a table in a cylinder and may be asked to lie still for up to 60 minutes at a time.

This study will not have a direct benefit for participants. However, knowledge gained may help researchers identify ways to improve movement in people with a brain injury, such as chronic stroke.

DETAILED DESCRIPTION:
Objectives

Non-invasive brain stimulation can modulate motor function in healthy volunteers and stroke patients when applied over the primary motor cortex (M1). M1 is an evident target for therapeutic interventions given its key role in motor control and learning. However, given the wide variety of motor dysfunctions following focal neurological injuries such as stroke, it is desirable to find out whether alternative neuronal structures could also be responsive to non-invasive brain stimulation for enhancing motor recovery. The cerebellum is an attractive target for therapeutic non-invasive brain stimulation since (i) the cerebellum plays a pivotal role in motor learning of reaching and movement synchronization tasks, (ii) the deep cerebellar nuclei are involved in the regulation of M1 neuronal activity through their excitatory drive to M1, and (iii) the cerebellum may be adaptively recruited after brain injury.

The purpose of this study is to find out if application of non-invasive transcranial DC stimulation (tDCS) can modulate motor cortical function. We hypothesize that tDCS of the cerebellar hemisphere ipsilateral (Cerebellum IPSI) to the target hand will modulate corticomotor excitability and motor function in healthy volunteers.

Study Population

40 healthy volunteers (18-40 years).

Design

This proof of principle study will determine if tDCS applied over the cerebellum can modulate focally motor excitability (as assessed by TMS) and motor performance. The stimulation parameters to be studied are polarity (anodal, cathodal and sham tDCS) and intensity (1 mA and 2 mA). The focality of stimulation will be addressed by applying tDCS over the neck and over M1 in separate control sessions, and by monitoring changes in cerebello-cortical excitability with paired-pulse TMS.

The outcome measures will be changes in motor cortical excitability as measured with TMS and in performance of an isometric pinch force task, a reaching task, and a motor sequence timing task. Attention and mood will be assessed to rule out nonspecific arousal effects. Paired-pulse TMS will be used to demonstrate modulations in cerebello-cortical connections and to characterize changes in intra-cortical excitability.

ELIGIBILITY:
* INCLUSION CRITERIA:
* age between 18-40 years
* able to perform tasks required by the study
* willing and able to give consent

EXCLUSION CRITERIA:

* unable to perform the tasks required by the study
* history of severe alcohol or drug abuse, psychiatric illness like severe depression, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score [MMSE] of 23 or less), or degenerative brain processes such as Alzheimer's disease
* severe uncontrolled medical problems (e.g., cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others), more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease
* problems with movement of the hands
* receiving drugs acting primarily on the central nervous system, which lower the seizure threshold, such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants (for the TMS component only)
* pregnant (for the MRI component only)
* medical or technical contraindications to MRI procedures or devices producing artifacts that impair MRI signal (e.g., pacemakers, implanted medication pumps, cochlear devices, neural stimulators, metal in the cranium, surgical clips, and other metal/magnetic implants, claustrophobia)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-12-14; Study Completion 2008-08-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Antal A, Nitsche MA, Kincses TZ, Kruse W, Hoffmann KP, Paulus W. Facilitation of visuo-motor learning by transcranial direct current stimulation of the motor and extrastriate visual areas in humans. Eur J Neurosci. 2004 May;19(10):2888-92. doi: 10.1111/j.1460-9568.2004.03367.x. PMID 15147322
- [Background] Khedr EM, Ahmed MA, Fathy N, Rothwell JC. Therapeutic trial of repetitive transcranial magnetic stimulation after acute ischemic stroke. Neurology. 2005 Aug 9;65(3):466-8. doi: 10.1212/01.wnl.0000173067.84247.36. PMID 16087918